CLINICAL TRIAL: NCT06347289
Title: Refusal of Organ Donation: a Study of Psychological, Anthropological and Cultural Factors
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Collaborators: Agence de La Biomédecine (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHSD_0024_REA
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Psychology; Anthropology; Refusal, Organ Donation
Keywords: refusal; organ donation; corpse; psychology; anthropology
MeSH Terms: conditions — Treatment Refusal; Cadaver

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Hospital of Saint Denis (HSD) has been involved for several years in the dynamics of organ donation. In spite of the evolution of the practices of coordination of the collection of samples, the rate of refusal of organ donation is increasing in our hospital, contrary to the rest of France.

Based on hypotheses derived from psychological and anthropological perspectives, this survey will provide first-hand information on the personal, family and cultural issues related to organ donation. It will be a question of identifying and locating individual and collective representations concerning death, its definition, and the associated symbols and rites. Based on the collection of these representations, we will be able to propose hypotheses of a psychological, social and anthropological nature on resistance to organ donation.

DETAILED DESCRIPTION:
The Hospital of Saint Denis (HSD) has been involved for several years in the dynamics of organ donation. In spite of the evolution of the practices of coordination of the collection of samples, the rate of refusal of organ donation is increasing in our hospital, contrary to the rest of France.

Based on hypotheses derived from psychological and anthropological perspectives, this survey will provide first-hand information on the personal, family and cultural issues related to organ donation. It will be a question of identifying and locating individual and collective representations concerning death, its definition, and the associated symbols and rites. Based on the collection of these representations, we will be able to propose hypotheses of a psychological, social and anthropological nature on resistance to organ donation.

Methodology :

Mixed quantitative and qualitative study

1. Questionnaire: The collection will be carried out prospectively on the hospital site for a period of 12 months. At the rate of one day per week. We estimate that we will be able to include 100 subjects during this period. Only those who have completed all the questionnaires will be included in the study. The collection will focus on the characteristics of the respondent (sex, age etc...) and will consist of 4 fields of questioning with open and closed questions (Biological and symbolic functioning associated with the organs that may be harvested, representation of death, fate of the corpse, and philosophical and religious positions regarding death and the corpse. Questions also on representations of the relationship between the hospital institution and the dead body: autopsy, brain death, organ removal, etc.)
2. Participant observation: by social science researcher. Targeted participation at key moments of the process leading to organ harvesting (medical staff in resuscitation, announcement interview, collection of non-opposition) allowing to carry out an ethnography. Duration: 3 months
3. Semi-structured interviews: at the end of the observation, concerning the various hospital actors in the organ donation process, both at the resuscitation level and the coordination of organ retrieval and the various professions (doctors, nurses, nursing auxiliaries). Number of interviews: 20

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the survey

Exclusion Criteria:

* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People and patients who visited Delafontaine's hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Demographic information | [day 1]
  Sex
Demographic information | [day 1]
  Age
Demographic information | [day 1]
  Nationality
Demographic information | [day 1]
  Mother tongue

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hopitalier de Saint-Denis, Saint-Denis, Seine Saint Denis, France